CLINICAL TRIAL: NCT02812511
Title: Pathophysiology Analysis of "Costello Syndrome" on Cellular Models
Acronym: COSTELLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2015/05
Record Dates: First submitted 2016-06-14; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Costello Syndrome
MeSH Terms: conditions — Costello Syndrome | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skin biopsy (Experimental)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Skin biopsy is performed at the arm with a punch of 3 mm in diameter or a scalpel under local anesthesia, and then preserved in low glucose DMEM at room temperature.

SUMMARY:
The objective is to collect skin biopsies rom patients with Costello syndrome to analyze the molecular mechanisms responsible for this syndrome caused by a mutation in the HRAS gene and the effects of this mutation on energy metabolism and mitochondrial physiology.

ELIGIBILITY:
Inclusion Criteria:

* Children aged over 2 years and under 18
* Children with a Costello Syndrome or Syndrome Cardio-Facio-Cutaneous

Exclusion Criteria:

* Previous history allergic to anesthetics

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Measurement of HRASG12V mutation on mitochondrial energy metabolism | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No